CLINICAL TRIAL: NCT03458988
Title: Pilot Study to Validate a Novel Blood-pressure Measuring Device in Patients Carrying a Left Ventricular Assist Device
Brief Title: Blood-pressure Measuring in Patients Carrying a Left Ventricular Assist Device
Acronym: LVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01570
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Left Ventricular Assist Device
Keywords: Blood pressure measuring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Nellcor™ Adult SpO2 Sensor
  Interventions: Device: Blood-pressure measuring (Nellcor™ Adult SpO2 Sensor)

INTERVENTIONS:
Device: Blood-pressure measuring (Nellcor™ Adult SpO2 Sensor) — Data will be acquired for 10 minutes with a reusable off the shelf adult SpO2 sensor. The Nellcor™ Adult SpO2 Sensor, model DS-100A, is indicated for use when continuous noninvasive arterial oxygen saturation and pulse rate monitoring are required for patients weighing greater than 40 kg.
  Other Names: Nellcor™ Adult SpO2 Sensor

SUMMARY:
To prove the novel device is able to reliably detect pulsatility in patients with CF-VADs and to analyze whether pre-programmed intrinsic pulsatility of the 3rd generation CF-VADs can also be picked up. The study is not designed to measure blood pressure.

Should this pilot study be successful in detecting enough pulsatility a follow-up study would then try to transfer the results into blood-pressure values with the help of comparators in order to identify an easier and more reliable method to measure BP in CF-VAD patients. .

DETAILED DESCRIPTION:
The number of patients supported by left ventricular assist device (LVAD) is increasing as durable mechanical support has become widely available for end stage heart failure as destination therapy and as bridge to transplantation. The accurate measurement of blood pressure (BP) as well as the recognition and management of hypertension in patients with LVADs is an essential component of optimal clinical care. Hypertension is an established long-term risk factor for cardiovascular disease. The measurement of BP and the management of hypertension in patients with CF-VADs can present unique challenges. Patients with LVADs often do not have a palpable pulse, and therefore traditional BP measurement by auscultation or automated cuff is less reliable. Conventional occlusive BP measurement is able to to pick up signals in approximately 50% of cases due to coincidental phases of pulsatility. The arterial line is the gold standard, but is an invasive procedure and not practical for routine outpatient use.

Although efforts are underway to identify an easier and more reliable method to measure ambulatory BP in these patients not one has been able to match the quality of an invasive arterial line.

ELIGIBILITY:
Inclusion Criteria:

* Patients carrying one of the two third generation CF-VADS (Heartware HVAD, Heartmate 3)
* Patients >18y
* Good understanding of written and oral German
* Signed informed consent
* Scheduled for routine outpatient appointment.

Exclusion Criteria:

* In the population of the outpatient clinic's CV-LVAD patients no known exclusion criteria exists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
RR (Riva Rocci, indirect blood pressure measurement) in LVAD | 10 min blood measuring
  Detect pulsatility in CF-VAD (Continuous flow- ventricular assist device) patients sufficient to calculate comprehensible blood-pressure values in future follow-up studies

CONTACTS AND LOCATIONS:
Overall Officials: David Reineke, MD, Principal Investigator — University Hospial Bern, Cardio Vascular Surgery
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Background] Saeed O, Jermyn R, Kargoli F, Madan S, Mannem S, Gunda S, Nucci C, Farooqui S, Hassan S, Mclarty A, Bloom M, Zolty R, Shin J, D'Alessandro D, Goldstein DJ, Patel SR. Blood pressure and adverse events during continuous flow left ventricular assist device support. Circ Heart Fail. 2015 May;8(3):551-6. doi: 10.1161/CIRCHEARTFAILURE.114.002000. Epub 2015 Apr 13. PMID 25870369
- [Background] Lampert BC, Eckert C, Weaver S, Scanlon A, Lockard K, Allen C, Kunz N, Bermudez C, Bhama JK, Shullo MA, Kormos RL, Dew MA, Teuteberg JJ. Blood pressure control in continuous flow left ventricular assist devices: efficacy and impact on adverse events. Ann Thorac Surg. 2014 Jan;97(1):139-46. doi: 10.1016/j.athoracsur.2013.07.069. Epub 2013 Sep 25. PMID 24075484